CLINICAL TRIAL: NCT03506100
Title: The Effects of Swimming and Swimming Complemented With Water Walking on Spirometry Values
Brief Title: The Effects of Water Walking on Spirometry Values
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Castelo Branco (Other)
Responsible Party: Principal Investigator, Pedro Alexandre Duarte Mendes, Principal Investigator, Instituto Politécnico de Castelo Branco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ESE IPCB_01
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Influence of Water Walking in Spirometric Values
Keywords: Spirometry; swimming; water walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- water walking in spirometric values (Other): Experimental: practice swimming complemented with water walking
  Interventions: Other: Water Walking

INTERVENTIONS:
Other: Water Walking — Practice swimming complemented with water walking at the end of each session and those who only practice swimming. In this study participated 28 subjects (mean age, 7.68 ± 1.16 years) and was divided into two groups: swimming group (SG) (N=9) and swimming complemented with water walking group (SWWG) (N=19). The study was performed in 12 weeks with 3 moments of evaluation (M1, M2 and M3) , with two sessions per week of 45 minutes each, we wanted to identify the benefits in pulmonary function - Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 second (FEV1) and Peak Expiratory Flow (PEF). The water walking activity occurred in the end of each session for 6 minutes, performed in straight line with the water level at the children's chest. The spirometry tests were realized with the microQuark Spirometer®.

SUMMARY:
The objective of this study was verify if there are differences in spirometry values in children aged between 6 and 12 years who practice swimming complemented with water walking at the end of each session and those who only practice swimming.

DETAILED DESCRIPTION:
Spirometry is a standard pulmonary function test that measures how an individual inhales or exhales volumes of air as a function time. It is the most important and most frequently performed pulmonary function testing procedure, having become indispensable for the prevention, diagnosis and evaluation of various respiratory impairments. However, there have been only a few studies addressing the effect of physical activity on pulmonary function test results and investigating the association between body composition and respiratory parameters in sports activities [1,2,3]. The objective of this study was verify if there are differences in spirometry values in children aged between 6 and 12 years who practice swimming complemented with water walking at the end of each session and those who only practice swimming. In this study participated 28 subjects (mean age, 7.68 ± 1.16 years) and was divided into two groups: swimming group (SG) (N=9) and swimming complemented with water walking group (SWWG) (N=19). The study was performed in 12 weeks with 3 moments of evaluation (M1, M2 and M3) , with two sessions per week of 45 minutes each, we wanted to identify the benefits in pulmonary function - Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 second (FEV1) and Peak Expiratory Flow (PEF). The water walking activity occurred in the end of each session for 6 minutes, performed in straight line with the water level at the children's chest. The spirometry tests were realized with the microQuark Spirometer®. For the analysis of the results, we used descriptive statistics, the Shapiro Wilk test for testing the normality of the sample and for the inferential statistics the Mann-Whitney tests, Friedman's Anova, and d-Cohen for the magnitude of effect.

ELIGIBILITY:
Inclusion Criteria:

* classes of the level of adaptation to the aquatic environment

Exclusion Criteria:

* Students who did not belong to this age group, that is, less than 6 years old or over 12, who attended classes only once a week, were athletes at a competitive level, and children with a 6 months and / or more than 12 months.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
spirometric values | 12 weeks
  The spirometry tests were realized with the microQuark Spirometer®.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Mendes, PhD, Principal Investigator — Instituto Politécnico de Castelo Branco

IPD SHARING:
Plan to Share IPD: Undecided